CLINICAL TRIAL: NCT04845620
Title: A Phase 3, 4-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-151 Cream 0.05% Administered QD in Subjects With Atopic Dermatitis
Brief Title: Trial of PDE4 Inhibition With Roflumilast for the Management of Atopic Dermatitis (Integument-PED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARQ-151-315
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roflumilast Cream 0.05% (Experimental): Participants applied roflumilast cream 0.05% qd for 4 weeks.
  Interventions: Drug: Roflumilast Cream 0.05%
- Vehicle Cream (Placebo Comparator): Participants applied vehicle cream qd for 4 weeks.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Roflumilast Cream 0.05% — Roflumilast cream for topical application.
  Other Names: ARQ-151
  Arms: Roflumilast Cream 0.05%
Drug: Vehicle Cream — Vehicle cream matched to roflumilast cream for topical application.
  Arms: Vehicle Cream

SUMMARY:
This was a Phase 3, 4-week, double-blind study to assess the safety and efficacy of ARQ-151 cream compared to vehicle cream applied once daily (qd) for 4 weeks in children 2 to 5 years of age with atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent by parent(s) or legal guardian as required by local laws.
2. Males and females, ages 2 to 5 years old at time of signing Informed Consent (Screening) and at Baseline (Day 1).
3. Diagnosed with atopic dermatitis for at least 6 weeks, as determined by the Investigator. Stable disease for the past 4 weeks with no significant flares in atopic dermatitis before screening.
4. In good health as judged by the Investigator.
5. Subjects considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

1. Subjects with any serious medical condition or clinically significant abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator
2. Has unstable AD or any consistent requirement for high potency topical steroids.
3. Subjects who are unwilling to refrain from prolonged sun exposure for 4 weeks prior to Baseline/Day 1 and during the study.
4. Previous treatment with ARQ-151.
5. Parent(s)/legal guardian(s) who are unable to communicate, read, or understand the local language(s). Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
6. Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members of enrolled (in other studies of ARQ-151) subjects living in the same house.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 652 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (76):
- United States (71):
  - Arcutis Clinical Site 56, Birmingham, Alabama
  - Arcutis Clinical Site 14, Birmingham, Alabama
  - Arcutis Clinical Site 69, Montgomery, Alabama
  - Arcutis Clinical Site 68, Gilbert, Arizona
  - Arcutis Clinical Site 26, Scottsdale, Arizona
  - Arcutis Clinical Site 50, Bryant, Arkansas
  - Arcutis Clinical Site 59, Fort Smith, Arkansas
  - Arcutis Clinical Site 71, Little Rock, Arkansas
  - Arcutis Clinical Site 09, Inglewood, California
  - Arcutis Clinical Site 45, Rancho Santa Margarita, California
  - Arcutis Clinical Site 30, San Diego, California
  - Arcutis Clinical Site 70, Thousand Oaks, California
  - Arcutis Clinical Site 48, Boca Raton, Florida
  - Arcutis Clinical Site 33, Coral Gables, Florida
  - Arcutis Clinical Site 12, Coral Gables, Florida
  - Arcutis Clinical Site 11, Delray Beach, Florida
  - Arcutis Clinical Site 28, Largo, Florida
  - Arcutis Clinical Site 79, Miami, Florida
  - Arcutis Clinical Site 43, Miami, Florida
  - Arcutis Clinical Site 10, Miami Lakes, Florida
  - Arcutis Clinical Site 35, North Miami Beach, Florida
  - Arcutis Clinical Site 75, Wellington, Florida
  - Arcutis Clinical Site 20, Sandy Springs, Georgia
  - Arcutis Clinical Site 82, Boise, Idaho
  - Arcutis Clinical Site 60, Chicago, Illinois
  - Arcutis Clinical Site 07, Rolling Meadows, Illinois
  - Arcutis Clinical Site 42, Clarksville, Indiana
  - Arcutis Clinical Site 21, Plainfield, Indiana
  - Arcutis Clinical Site 57, West Lafayette, Indiana
  - Arcutis Clinical Site 22, Louisville, Kentucky
  - Arcutis Clinical Site 46, Louisville, Kentucky
  - Arcutis Clinical Site 84, Baton Rouge, Louisiana
  - Arcutis Clinical Site 34, Lake Charles, Louisiana
  - Arcutis Clinical Site 51, Metairie, Louisiana
  - Arcutis Clinical Site 40, Metairie, Louisiana
  - Arcutis Clinical Site 77, Columbia, Maryland
  - Arcutis Clinical Site 13, Rockville, Maryland
  - Arcutis Clinical Site 15, Rockville, Maryland
  - Arcutis Clinical Site 53, Auburn Hills, Michigan
  - Arcutis Clinical Site 41, Bay City, Michigan
  - Arcutis Clinical Site 36, Clarkston, Michigan
  - Arcutis Clinical Site 72, Troy, Michigan
  - Arcutis Clinical Site 05, New Brighton, Minnesota
  - Arcutis Clinical Site 47, Saint Joseph, Missouri
  - Arcutis Clinical Site 16, Reno, Nevada
  - Arcutis Clinical Site 55, Lebanon, New Hampshire
  - Arcutis Clinical Site 54, Brooklyn, New York
  - Arcutis Clinical Site 44, New York, New York
  - Arcutis Clinical Site 32, Rochester, New York
  - Arcutis Clinical Site 58, Cincinnati, Ohio
  - Arcutis Clinical Site 81, Mason, Ohio
  - Arcutis Clinical Site 01, Gresham, Oregon
  - Arcutis Clinical Site 52, Portland, Oregon
  - Arcutis Clinical Site 63, Portland, Oregon
  - Arcutis Clinical Site 65, Bethlehem, Pennsylvania
  - Arcutis Clinical Site 31, Hershey, Pennsylvania
  - Arcutis Clinical Site 24, Newtown Square, Pennsylvania
  - Arcutis Clinical Site 62, Charleston, South Carolina
  - Arcutis Clinical Site 39, Summerville, South Carolina
  - Arcutis Clinical Site 08, Austin, Texas
  - Arcutis Clinical Site 27, Bellaire, Texas
  - Arcutis Clinical Site 74, Fort Worth, Texas
  - Arcutis Clinical Site 66, Frisco, Texas
  - Arcutis Clinical Site 61, Grapevine, Texas
  - Arcutis Clinical Site 04, Houston, Texas
  - Arcutis Clinical Site 02, San Antonio, Texas
  - Arcutis Clinical Site 18, San Antonio, Texas
  - Arcutis Clinical Site 03, South Jordan, Utah
  - Arcutis Clinical Site 06, Burke, Virginia
  - Arcutis Clinical Site 76, Charlottesville, Virginia
  - Arcutis Clinical Site 25, Spokane, Washington
- Canada (5):
  - Arcutis Clinical Site 29, Calgary, Alberta
  - Arcutis Clinical Site 64, Winnipeg, Manitoba
  - Arcutis Clinical Site 73, Burlington, Ontario
  - Arcutis Clinical Site 36, Markham, Ontario
  - Arcutis Clinical Site 78, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Eichenfield LF, Serrao R, Prajapati VH, Browning JC, Swanson L, Funk T, Gonzalez ME, Hebert AA, Lee M, Boguniewicz M, Simpson EL, Seal MS, Krupa D, Hanna D, Snyder S, Burnett P, Chu DH, Almaraz E, Higham RC, Berk DR. Efficacy and Safety of Once-Daily Roflumilast Cream 0.05% in Pediatric Patients Aged 2-5 Years With Mild-to-Moderate Atopic Dermatitis (INTEGUMENT-PED): A Phase 3 Randomized Controlled Trial. Pediatr Dermatol. 2025 Mar-Apr;42(2):296-304. doi: 10.1111/pde.15840. Epub 2025 Feb 20. PMID 39980188

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 109 centers in the United States, Canada, and Poland.
Period: Overall Study
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Started | 437 | 215
Completed | 410 | 192
Not Completed | 27 | 23
Not completed — Withdrawal by Subject | 11 | 10
Not completed — Adverse Event | 5 | 4
Not completed — Lost to Follow-up | 5 | 4
Not completed — Lack of Efficacy | 4 | 4
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream | Total
Number analyzed (Participants) | 437 | 215 | 652
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.3 (1.09) | 3.2 (1.10) | 3.3 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 99 | 310
  Male | 226 | 116 | 342
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 82 | 31 | 113
  Not Hispanic or Latino | 352 | 184 | 536
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 37 | 17 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 68 | 32 | 100
  White | 295 | 156 | 451
  More than one race | 28 | 4 | 32
  Unknown or Not Reported | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Success at Week 4
Description: The percentage of participants with vIGA-AD success at Week 4 is presented. The vIGA-AD is a static evaluation of qualitative overall AD severity with five severity grades (reported as score of 0 'clear' to 4 'severe' with higher scores indicating greater symptom severity. vIGA success was defined as score of 'clear' or 'almost clear' plus a 2-grade improvement from baseline.
Time Frame: Week 4
Population: All randomized participants are included, 1 participant in the Roflumilast Cream 0.05% arm was inadvertently treated prior to randomization and thus excluded from analysis.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Number analyzed (Participants) | 436 | 215
percentage of participants | 25.4 [20.95 to 30.34] | 10.7 [6.77 to 16.45]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; vIGA Success at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by randomized baseline vIGA-AD with multiple imputation of missing observations; Odds Ratio (OR) = 2.89, 97.5% CI 2-sided [1.648 to 5.064] — Stratified by randomized baseline vIGA-AD with multiple imputation of missing observations

2. Secondary Outcome: Achievement of vIGA-AD Success at Week 4 in Participants With 'Moderate' Baseline vIGA-AD
Description: The percentage of participants with vIGA-AD success at Week 4 who had 'moderate' vIGA-AD score (vIGA score of 3) at baseline is presented. The vIGA-AD is a static evaluation of qualitative overall AD severity with five severity grades (reported as score of 0 'clear' to 4 'severe' with higher scores indicating greater symptom severity. vIGA-AD success was defined as score of 'clear' or 'almost clear' plus a 2-grade improvement from baseline in participants with moderate vIGA-AD baseline.
Time Frame: Week 4
Population: All randomized participants with a baseline vIGA score of 'moderate' are included.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Number analyzed (Participants) | 333 | 171
percentage of participants | 27.7 [22.55 to 33.62] | 11.0 [6.67 to 17.73]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; vIGA Success at Week 4 in Participants with Moderate Baseline vIGA; Test type: Superiority; p < 0.0001, Chi-squared; Multiple imputation of missing observations; Odds Ratio (OR) = 3.10, 97.5% CI 2-sided [1.662 to 5.772] — Multiple imputation of missing observations

3. Secondary Outcome: Achievement of 75% Reduction in the Eczema Area and Severity Index (EASI-75) at Week 4 In Participants With 'Moderate' Baseline vIGA
Description: The percentage of participants with a moderate baseline vIGA-AD score who achieved EASI-75 is presented. EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head {10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Time Frame: Week 4
Population: All randomized participants are included, with the exception of 1 participant in the Roflumilast Cream 0.05% arm who was inadvertently treated prior to randomization and thus excluded from analysis.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Number analyzed (Participants) | 436 | 215
percentage of participants | 39.4 [34.21 to 44.81] | 20.6 [15.06 to 27.55]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; EASI-75 at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by randomized baseline vIGA-AD with multiple imputation of missing observations; Odds Ratio (OR) = 2.47, 97.5% CI 2-sided [1.578 to 3.870] — Stratified by randomized baseline vIGA-AD with multiple imputation of missing observations

4. Secondary Outcome: Achievement of vIGA-AD Score of 'Clear' or 'Almost Clear'
Description: The percentage of participants with vIGA-AD score of 'clear' or 'almost clear' at Week 4 is presented. The vIGA is a static evaluation of qualitative overall AD severity with five severity grades (reported as score of 0 'clear' to 4 'severe' with higher scores indicating greater symptom severity.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Number analyzed (Participants) | 436 | 215
percentage of participants | 35.4 [30.39 to 40.66] | 14.6 [9.94 to 20.86]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; vIGA Score of 'Clear' or 'Almost Clear' at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by randomized baseline vIGA-AD with multiple imputation of missing observations; Odds Ratio (OR) = 3.29, 97.5% CI 2-sided [1.980 to 5.475] — Stratified by randomized baseline vIGA-AD with multiple imputation of missing observations

5. Secondary Outcome: Achievement of vIGA-AD Success at Week 2
Description: The percentage of participants with vIGA-AD success at Week 2 is presented. The vIGA-AD is a static evaluation of qualitative overall AD severity with five severity grades (reported as score of 0 'clear' to 4 'severe' with higher scores indicating greater symptom severity. vIGA success was defined as score of 'clear' or 'almost clear' plus a 2-grade improvement from baseline.
Time Frame: Week 2
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Number analyzed (Participants) | 436 | 215
percentage of participants | 21.2 [17.13 to 25.98] | 6.8 [3.85 to 11.88]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by baseline vIGA-AD with multiple imputation of missing observations; Odds Ratio (OR) = 3.74, 97.5% CI 2-sided [1.912 to 7.313] — Stratified by baseline vIGA-AD with multiple imputation of missing observations

6. Secondary Outcome: Achievement of vIGA-AD Success at Week 1
Description: The percentage of participants with vIGA-AD success at Week 1 is presented. The vIGA-AD is a static evaluation of qualitative overall AD severity with five severity grades (reported as score of 0 'clear' to 4 'severe' with higher scores indicating greater symptom severity. vIGA-AD success was defined as score of 'clear' or 'almost clear' plus a 2-grade improvement from baseline.
Time Frame: Week 1
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Number analyzed (Participants) | 436 | 215
percentage of participants | 9.4 [6.72 to 13.02] | 0.9 [0.22 to 3.88]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; vIGA-AD Success at Week 1; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by randomized baseline vIGA-AD with multiple imputation of missing data; Odds Ratio (OR) = 11.44, 97.5% CI 2-sided [2.216 to 59.101] — Stratified by randomized baseline vIGA-AD with multiple imputation of missing data

7. Secondary Outcome: Achievement of vIGA-AD of 'Clear' or 'Almost Clear' at Week 2
Description: The percentage of participants with vIGA-AD score of 'clear' or 'almost clear' at Week 2 is presented. The vIGA-AD is a static evaluation of qualitative overall AD severity with five severity grades (reported as score of 0 'clear' to 4 'severe' with higher scores indicating greater symptom severity.
Time Frame: Week 2
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Number analyzed (Participants) | 436 | 215
percentage of participants | 30.4 [25.67 to 35.58] | 10.6 [6.74 to 16.42]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; vIGA-AD of Clear or Almost Clear at Week 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by randomized baseline vIGA-AD with multiple imputation of missing data; Odds Ratio (OR) = 3.80, 97.5% CI 2-sided [2.137 to 6.761] — Stratified by randomized baseline vIGA-AD with multiple imputation of missing data

8. Secondary Outcome: Achievement of vIGA-AD of 'Clear' or 'Almost Clear' at Week 1
Description: The percentage of participants with vIGA-AD score of 'clear' or 'almost clear' at Week 1 is presented. The vIGA-AD is a static evaluation of qualitative overall AD severity with five severity grades (reported as score of 0 'clear' to 4 'severe' with higher scores indicating greater symptom severity.
Time Frame: Week 1
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
Number analyzed (Participants) | 436 | 215
percentage of participants | 17.00 [13.32 to 21.37] | 3.7 [1.73 to 7.83]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; vIGA-AD of Clear or Almost Clear at Week 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by baseline vIGA-AD with multiple imputation of missing data; Odds Ratio (OR) = 5.75, 97.5% CI 2-sided [2.342 to 14.113] — Stratified by baseline vIGA-AD with multiple imputation of missing data

ADVERSE EVENTS:
Time Frame: Up to ~6 weeks
Arm/Group | Roflumilast Cream 0.05% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/437 | 0/215
Serious Adverse Events (participants affected / at risk) | 1/437 | 0/215
Other Adverse Events (participants affected / at risk) | 0/437 | 0/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Cream 0.05% (N=437) | Vehicle Cream (N=215)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT04845620/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT04845620/SAP_001.pdf